CLINICAL TRIAL: NCT03904108
Title: Phase-II Trial of Platinum-Based Chemotherapy Plus Ramucirumab in Patients With Advanced NSCLC Who Have Progressed on First Line Anti-PD-1 Immunotherapy
Brief Title: Platinum-Based Chemotherapy Plus Ramucirumab in Patients With Advanced NSCLC Who Have Progressed on First Line Anti-PD-1 Immunotherapy
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: insufficient patient population to complete trial as planned
Sponsor: ROGER S KERESZTES MD (Other)
Responsible Party: Sponsor-Investigator, ROGER S KERESZTES MD, Clinical Associate Professor, Stony Brook University
Organization: Stony Brook University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB2019-00094
Record Dates: First submitted 2019-04-02; First posted 2019-04-04 (Actual); Results first posted 2022-05-26 (Actual); Last update posted 2022-05-26 (Actual); Status verified 2022-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: NSCLC; Immunotherapy; Ramucirumab; anti-PD-1
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Ramucirumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Ramucirumab (Experimental): Ramucirumab 10 mg/kg IV day 1, every 3 weeks for 4 cycles
  Interventions: Drug: Ramucirumab

INTERVENTIONS:
Drug: Ramucirumab — platinum doublets chemotherapy plus ramucirumab, intravenously(IV)
  Other Names: cyramza; BLA 125477

SUMMARY:
This is a non-randomized, phase-II study of platinum doublet chemotherapy plus ramucirumab in patients with advanced NSCLC who have progressed on first line anti-PD-1 Immunotherapy. Up to 25 evaluable participants will be enrolled over a period of 2 years. Seven patients will be recruited at the first stage .Eligible patients would include those treated with a PD-1 inhibitor as primary therapy and exhibit evidence of disease progression, but maintain a good performance status.

The investigators hypothesize that immune therapy acts as chemo-sensitizer and patients treated with standard platinum-based combination chemotherapy with the addition of the anti-angiogenic agent Ramucirumab, after immunotherapy will have higher response rates

DETAILED DESCRIPTION:
OBJECTIVES:

Primary Objective

1. To assess the objective response rate to a three-drug regimen (a platinum doublet plus an anti-angiogenic agent) in patients with non-small cell lung cancer who fail to respond, or progress after an initial response, to primary therapy with an immune checkpoint inhibitor.
2. To assess the toxicity profile of the three-drug regimen in this population compared to historical treatment-naïve population (as published in literature)

Exploratory Objective

1. To investigate the role of peripheral blood CD 8+ T cells, absolute eosinophil count (AEC) and circulating tumor cells (CTC) as biomarkers of response to salvage chemotherapy after primary immunotherapy
2. To investigate the role of plasma carbonic anhydrase IX level as predictive biomarker of response to ramucirumab.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed stage IV NSCLC per 8th IASCL (International Association for the Study of Lung Cancer) of squamous and non-squamous histology, with progression on first line anti-PD1 immunotherapy.
2. Oligo-metastatic stage IV patients who received concurrent chemotherapy with thoracic radiation, followed by durvalumab consolidation and had progression of disease.
3. Locally advanced un-resectable NSCLC patients who received concurrent chemotherapy with thoracic radiation, followed by durvalumab consolidation and had progression of disease.
4. Males or females at least 18 years of age.
5. ECOG (Eastern Cooperative Oncology Group) performance status of 0 or 1.
6. Measureable disease by CT or MRI per RECIST 1.1 criteria.
7. Life expectancy of at least 3 months.
8. Resolution of all clinically significant toxic effects of prior anticancer therapy to Grade ≤1 by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE), Version 4.0.
9. The participant must have adequate organ function, defined as:

   * Total bilirubin less than or equal to the upper limit of normal value (ULN), aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤2.5 x ULN, or ≤5 x ULN if the transferase elevation was due to liver metastases.
   * Serum creatinine ≤1.5 x ULN or calculated creatinine clearance ≥50 mL/min (per the Cockcroft-Gault formula or equivalent and/or 24-hour urine collection [Cockcroft-Gault glomerular filtration rate = (140-age) * (Wt in kg) * (0.85 if female) / (72 * Cr) where "Cr" is serum creatinine]).
   * Absolute neutrophil count (ANC) ≥1.5 x 103/μL (≥1.5 x 109/L), hemoglobin ≥10.0 g/dL (≥ 6.2 mmol/L), and platelets ≥100 x 103/μL (≥100 x 109/L).
   * International Normalized Ratio (INR) less than or equal to 1.5, or prothrombin time and partial thromboplastin time less than or equal to 1.5 x ULN.
   * The participant does not have cirrhosis at a level of Child-Pugh B (or worse) or cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites resulting from cirrhosis and requiring ongoing treatment with diuretics and/or paracentesis.
10. Urinary protein is ≤1+ on dipstick or routine urinalysis (UA). If urine dipstick or routine analysis indicated proteinuria ≥2+, then a 24-hour urine must be collected and must demonstrate <1000 mg of protein in 24 hours to allow participation in the study.
11. Female subjects must have a negative urine or serum pregnancy test at screening (within 72 hours of first dose of study medication) if of childbearing potential or be of non-child bearing potential.
12. If of childbearing potential, female subjects must be willing to use two adequate barrier methods throughout the study, starting with the screening visit through 180 days after last dose of chemotherapeutic agents.

    Note: Abstinence is acceptable if this is the established and preferred contraception.
13. Male subjects with a female partner(s) of child-bearing potential must agree to use two adequate barrier methods throughout the trial starting with the screening visit through 180 days after the last dose of chemotherapy. Males with pregnant partners must agree to use a condom; no additional method of contraception is required for the pregnant partner.
14. The participant has voluntarily agreed to participate by giving written informed consent for the trial.

Exclusion Criteria:

1. Participant has received prior cytotoxic therapy or targeted oral agents for the treatment of their stage IV NSCLC. Participants with oligo-metastatic stage IV disease who received concurrent chemotherapy with thoracic radiation, followed by durvalumab consolidation with disease progression were eligible.
2. Participant has an EGFR (epidermal growth factor receptor) sensitizing mutation, ALK translocation and/or an ROS-1 gene rearrangement.
3. Participant has undergone major surgery within 28 days prior to screening, or subcutaneous venous access device placement within 7 days prior to screening. Furthermore, any partcipant with postoperative bleeding complications or wound complications from a surgical procedure performed in the last 2 months will be excluded.
4. Participant has untreated CNS (central nervous system) metastases. Participants with treated brain metastases were eligible if they were clinically stable with regard to neurologic function, off steroids after cranial irradiation (whole brain radiation therapy, focal radiation therapy, and stereotactic radiosurgery) ending at least 2 weeks prior to screening, or after surgical resection performed at least 28 days prior to screening. No evidence of Grade ≥1 CNS hemorrhage based on pretreatment MRI or IV contrast CT scan (performed within 21 days before screening).
5. There is radiologically documented evidence of major blood vessel invasion or encasement by cancer.
6. There is radiographic evidence of intra-tumor cavitation, regardless of tumor histology.
7. Participant has a history of uncontrolled hereditary or acquired thrombotic disorder.
8. Participant has a history of gross hemoptysis (defined as bright red blood or ≥1/2 teaspoon) within 2months prior to screening.
9. Participant has clinically relevant congestive heart failure (CHF; NYHA II-IV) or symptomatic or poorly controlled cardiac arrhythmia.
10. Participant has experienced any arterial thrombotic event, including myocardial infarction, unstable angina, cerebrovascular accident, or transient ischemic attack, within 6 months prior to screening.
11. Participant has uncontrolled arterial hypertension ≥150 / ≥90 mm Hg despite standard medical management.
12. Participant has a serious or non-healing wound, ulcer, or bone fracture within 28 days prior to screening.
13. Participant has significant bleeding disorders, vasculitis, or experienced Grade 3-4 gastrointestinal (GI) bleeding within 3 months prior to screening.
14. History of GI perforation and/or fistulae within 6 months prior to screening.
15. Participant has bowel obstruction,history or presence of inflammatory enteropathy or extensive intestinal resection (hemicolectomy or extensive small intestine resection with chronic diarrhea), Crohn's disease, ulcerative colitis, or chronic diarrhea.
16. Participant has peripheral neuropathy ≥Grade 2 (NCI-CTCAE v 4.0).
17. Participant has a serious illness or medical condition(s) including, but not limited to, the following:

    * Known human immunodeficiency virus (HIV) infection or acquired immunodeficiency syndrome (AIDS)-related illness.
    * Active or uncontrolled clinically serious infection.
    * Previous or concurrent malignancy except for basal or squamous cell skin cancer and/or in situ carcinoma of the cervix, or other solid tumours treated curatively and without evidence of recurrence for at least 3 years prior to screening.
    * Uncontrolled metabolic disorders or other nonmalignant organ or systemic diseases or secondary effects of cancer that induced a high medical risk and/or made assessment of survival uncertain.
    * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that might increase the risk associated with study participation or study drug administration, or might interfere with the interpretation of study results, and in the judgment of the investigator made the patient ineligible for entry into this study.
    * Participant has significant third-space fluid retention (for example, ascites or pleural effusion), and is not amenable for required repeated drainage.
    * Known allergy or hypersensitivity reaction to any of the treatment components.
    * Participant has a known history of active drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2019-06-27 (Actual); Primary Completion 2020-07-27 (Actual); Study Completion 2020-07-27 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Stony Brook University, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Siegel RL, Miller KD, Jemal A. Cancer Statistics, 2017. CA Cancer J Clin. 2017 Jan;67(1):7-30. doi: 10.3322/caac.21387. Epub 2017 Jan 5. PMID 28055103
- [Background] Schiller JH, Harrington D, Belani CP, Langer C, Sandler A, Krook J, Zhu J, Johnson DH; Eastern Cooperative Oncology Group. Comparison of four chemotherapy regimens for advanced non-small-cell lung cancer. N Engl J Med. 2002 Jan 10;346(2):92-8. doi: 10.1056/NEJMoa011954. PMID 11784875
- [Background] Sandler A, Gray R, Perry MC, Brahmer J, Schiller JH, Dowlati A, Lilenbaum R, Johnson DH. Paclitaxel-carboplatin alone or with bevacizumab for non-small-cell lung cancer. N Engl J Med. 2006 Dec 14;355(24):2542-50. doi: 10.1056/NEJMoa061884. PMID 17167137
- [Background] Sandler AB, Schiller JH, Gray R, Dimery I, Brahmer J, Samant M, Wang LI, Johnson DH. Retrospective evaluation of the clinical and radiographic risk factors associated with severe pulmonary hemorrhage in first-line advanced, unresectable non-small-cell lung cancer treated with Carboplatin and Paclitaxel plus bevacizumab. J Clin Oncol. 2009 Mar 20;27(9):1405-12. doi: 10.1200/JCO.2008.16.2412. Epub 2009 Feb 17. PMID 19224857
- [Background] Ramalingam SS, Dahlberg SE, Langer CJ, Gray R, Belani CP, Brahmer JR, Sandler AB, Schiller JH, Johnson DH; Eastern Cooperative Oncology Group. Outcomes for elderly, advanced-stage non small-cell lung cancer patients treated with bevacizumab in combination with carboplatin and paclitaxel: analysis of Eastern Cooperative Oncology Group Trial 4599. J Clin Oncol. 2008 Jan 1;26(1):60-5. doi: 10.1200/JCO.2007.13.1144. PMID 18165641
- [Background] Garon EB, Ciuleanu TE, Arrieta O, Prabhash K, Syrigos KN, Goksel T, Park K, Gorbunova V, Kowalyszyn RD, Pikiel J, Czyzewicz G, Orlov SV, Lewanski CR, Thomas M, Bidoli P, Dakhil S, Gans S, Kim JH, Grigorescu A, Karaseva N, Reck M, Cappuzzo F, Alexandris E, Sashegyi A, Yurasov S, Perol M. Ramucirumab plus docetaxel versus placebo plus docetaxel for second-line treatment of stage IV non-small-cell lung cancer after disease progression on platinum-based therapy (REVEL): a multicentre, double-blind, randomised phase 3 trial. Lancet. 2014 Aug 23;384(9944):665-73. doi: 10.1016/S0140-6736(14)60845-X. Epub 2014 Jun 2. PMID 24933332
- [Background] Camidge DR, Berge EM, Doebele RC, Ballas MS, Jahan T, Haigentz M Jr, Hoffman D, Spicer J, West H, Lee P, Yang L, Joshi A, Gao L, Yurasov S, Mita A. A phase II, open-label study of ramucirumab in combination with paclitaxel and carboplatin as first-line therapy in patients with stage IIIB/IV non-small-cell lung cancer. J Thorac Oncol. 2014 Oct;9(10):1532-9. doi: 10.1097/JTO.0000000000000273. PMID 25170639
- [Background] Doebele RC, Spigel D, Tehfe M, Thomas S, Reck M, Verma S, Eakle J, Bustin F, Goldschmidt J Jr, Cao D, Alexandris E, Yurasov S, Camidge DR, Bonomi P. Phase 2, randomized, open-label study of ramucirumab in combination with first-line pemetrexed and platinum chemotherapy in patients with nonsquamous, advanced/metastatic non-small cell lung cancer. Cancer. 2015 Mar 15;121(6):883-92. doi: 10.1002/cncr.29132. Epub 2014 Nov 6. PMID 25377507
- [Background] Brahmer J, Reckamp KL, Baas P, Crino L, Eberhardt WE, Poddubskaya E, Antonia S, Pluzanski A, Vokes EE, Holgado E, Waterhouse D, Ready N, Gainor J, Aren Frontera O, Havel L, Steins M, Garassino MC, Aerts JG, Domine M, Paz-Ares L, Reck M, Baudelet C, Harbison CT, Lestini B, Spigel DR. Nivolumab versus Docetaxel in Advanced Squamous-Cell Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Jul 9;373(2):123-35. doi: 10.1056/NEJMoa1504627. Epub 2015 May 31. PMID 26028407
- [Background] Borghaei H, Paz-Ares L, Horn L, Spigel DR, Steins M, Ready NE, Chow LQ, Vokes EE, Felip E, Holgado E, Barlesi F, Kohlhaufl M, Arrieta O, Burgio MA, Fayette J, Lena H, Poddubskaya E, Gerber DE, Gettinger SN, Rudin CM, Rizvi N, Crino L, Blumenschein GR Jr, Antonia SJ, Dorange C, Harbison CT, Graf Finckenstein F, Brahmer JR. Nivolumab versus Docetaxel in Advanced Nonsquamous Non-Small-Cell Lung Cancer. N Engl J Med. 2015 Oct 22;373(17):1627-39. doi: 10.1056/NEJMoa1507643. Epub 2015 Sep 27. PMID 26412456
- [Background] Herbst RS, Baas P, Kim DW, Felip E, Perez-Gracia JL, Han JY, Molina J, Kim JH, Arvis CD, Ahn MJ, Majem M, Fidler MJ, de Castro G Jr, Garrido M, Lubiniecki GM, Shentu Y, Im E, Dolled-Filhart M, Garon EB. Pembrolizumab versus docetaxel for previously treated, PD-L1-positive, advanced non-small-cell lung cancer (KEYNOTE-010): a randomised controlled trial. Lancet. 2016 Apr 9;387(10027):1540-1550. doi: 10.1016/S0140-6736(15)01281-7. Epub 2015 Dec 19. PMID 26712084
- [Background] Rittmeyer A, Barlesi F, Waterkamp D, Park K, Ciardiello F, von Pawel J, Gadgeel SM, Hida T, Kowalski DM, Dols MC, Cortinovis DL, Leach J, Polikoff J, Barrios C, Kabbinavar F, Frontera OA, De Marinis F, Turna H, Lee JS, Ballinger M, Kowanetz M, He P, Chen DS, Sandler A, Gandara DR; OAK Study Group. Atezolizumab versus docetaxel in patients with previously treated non-small-cell lung cancer (OAK): a phase 3, open-label, multicentre randomised controlled trial. Lancet. 2017 Jan 21;389(10066):255-265. doi: 10.1016/S0140-6736(16)32517-X. Epub 2016 Dec 13. PMID 27979383
- [Background] Reck M, Rodriguez-Abreu D, Robinson AG, Hui R, Csoszi T, Fulop A, Gottfried M, Peled N, Tafreshi A, Cuffe S, O'Brien M, Rao S, Hotta K, Leiby MA, Lubiniecki GM, Shentu Y, Rangwala R, Brahmer JR; KEYNOTE-024 Investigators. Pembrolizumab versus Chemotherapy for PD-L1-Positive Non-Small-Cell Lung Cancer. N Engl J Med. 2016 Nov 10;375(19):1823-1833. doi: 10.1056/NEJMoa1606774. Epub 2016 Oct 8. PMID 27718847
- [Background] Langer CJ, Gadgeel SM, Borghaei H, Papadimitrakopoulou VA, Patnaik A, Powell SF, Gentzler RD, Martins RG, Stevenson JP, Jalal SI, Panwalkar A, Yang JC, Gubens M, Sequist LV, Awad MM, Fiore J, Ge Y, Raftopoulos H, Gandhi L; KEYNOTE-021 investigators. Carboplatin and pemetrexed with or without pembrolizumab for advanced, non-squamous non-small-cell lung cancer: a randomised, phase 2 cohort of the open-label KEYNOTE-021 study. Lancet Oncol. 2016 Nov;17(11):1497-1508. doi: 10.1016/S1470-2045(16)30498-3. Epub 2016 Oct 10. PMID 27745820
- [Background] Antonia SJ, Villegas A, Daniel D, Vicente D, Murakami S, Hui R, Yokoi T, Chiappori A, Lee KH, de Wit M, Cho BC, Bourhaba M, Quantin X, Tokito T, Mekhail T, Planchard D, Kim YC, Karapetis CS, Hiret S, Ostoros G, Kubota K, Gray JE, Paz-Ares L, de Castro Carpeno J, Wadsworth C, Melillo G, Jiang H, Huang Y, Dennis PA, Ozguroglu M; PACIFIC Investigators. Durvalumab after Chemoradiotherapy in Stage III Non-Small-Cell Lung Cancer. N Engl J Med. 2017 Nov 16;377(20):1919-1929. doi: 10.1056/NEJMoa1709937. Epub 2017 Sep 8. PMID 28885881
- [Background] Patel JD, Socinski MA, Garon EB, Reynolds CH, Spigel DR, Olsen MR, Hermann RC, Jotte RM, Beck T, Richards DA, Guba SC, Liu J, Frimodt-Moller B, John WJ, Obasaju CK, Pennella EJ, Bonomi P, Govindan R. PointBreak: a randomized phase III study of pemetrexed plus carboplatin and bevacizumab followed by maintenance pemetrexed and bevacizumab versus paclitaxel plus carboplatin and bevacizumab followed by maintenance bevacizumab in patients with stage IIIB or IV nonsquamous non-small-cell lung cancer. J Clin Oncol. 2013 Dec 1;31(34):4349-57. doi: 10.1200/JCO.2012.47.9626. Epub 2013 Oct 21. PMID 24145346
- [Background] Radfar S, Wang Y, Khong HT. Activated CD4+ T cells dramatically enhance chemotherapeutic tumor responses in vitro and in vivo. J Immunol. 2009 Nov 15;183(10):6800-7. doi: 10.4049/jimmunol.0901747. Epub 2009 Oct 21. PMID 19846868
- [Background] Chen G, Emens LA. Chemoimmunotherapy: reengineering tumor immunity. Cancer Immunol Immunother. 2013 Feb;62(2):203-16. doi: 10.1007/s00262-012-1388-0. Epub 2013 Feb 7. PMID 23389507
- [Background] Fridlender ZG, Sun J, Singhal S, Kapoor V, Cheng G, Suzuki E, Albelda SM. Chemotherapy delivered after viral immunogene therapy augments antitumor efficacy via multiple immune-mediated mechanisms. Mol Ther. 2010 Nov;18(11):1947-59. doi: 10.1038/mt.2010.159. Epub 2010 Aug 3. PMID 20683443
- [Background] Schvartsman G, Peng SA, Bis G, Lee JJ, Benveniste MFK, Zhang J, Roarty EB, Lacerda L, Swisher S, Heymach JV, Fossella FV, William WN. Response rates to single-agent chemotherapy after exposure to immune checkpoint inhibitors in advanced non-small cell lung cancer. Lung Cancer. 2017 Oct;112:90-95. doi: 10.1016/j.lungcan.2017.07.034. Epub 2017 Aug 3. PMID 29191606
- [Background] Park SE, Lee SH, Ahn JS, Ahn MJ, Park K, Sun JM. Increased Response Rates to Salvage Chemotherapy Administered after PD-1/PD-L1 Inhibitors in Patients with Non-Small Cell Lung Cancer. J Thorac Oncol. 2018 Jan;13(1):106-111. doi: 10.1016/j.jtho.2017.10.011. Epub 2017 Oct 31. PMID 29101058
- [Background] Kamphorst AO, Pillai RN, Yang S, Nasti TH, Akondy RS, Wieland A, Sica GL, Yu K, Koenig L, Patel NT, Behera M, Wu H, McCausland M, Chen Z, Zhang C, Khuri FR, Owonikoko TK, Ahmed R, Ramalingam SS. Proliferation of PD-1+ CD8 T cells in peripheral blood after PD-1-targeted therapy in lung cancer patients. Proc Natl Acad Sci U S A. 2017 May 9;114(19):4993-4998. doi: 10.1073/pnas.1705327114. Epub 2017 Apr 26. PMID 28446615
- [Background] Stewart GD, O'Mahony FC, Laird A, Rashid S, Martin SA, Eory L, Lubbock AL, Nanda J, O'Donnell M, Mackay A, Mullen P, McNeill SA, Riddick AC, Aitchison M, Berney D, Bex A, Overton IM, Harrison DJ, Powles T. Carbonic anhydrase 9 expression increases with vascular endothelial growth factor-targeted therapy and is predictive of outcome in metastatic clear cell renal cancer. Eur Urol. 2014 Nov;66(5):956-63. doi: 10.1016/j.eururo.2014.04.007. Epub 2014 May 10. PMID 24821582
- [Background] Brown-Glaberman U, Marron M, Chalasani P, Livingston R, Iannone M, Specht J, Stopeck AT. Circulating Carbonic Anhydrase IX and Antiangiogenic Therapy in Breast Cancer. Dis Markers. 2016;2016:9810383. doi: 10.1155/2016/9810383. Epub 2016 Jan 28. PMID 26941473

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ramucirumab
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Ramucirumab
Number analyzed (Participants) | 3
Age, Customized [Number; unit: participants]
  Age Range 58-66 years | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  white,non-Hispanic | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Objective Response Per RECIST 1.1 as Assessed by Central Imaging
Description: Objective response (OR) is the occurrence of CR or PR as the best overall response. OR will be based on responses confirmed using the subsequent 6-weekly scan. OR is based on the Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: ≥18 weeks, up to maximum of 12 months
Population: Data were not collected
Arm/Group | Ramucirumab
Number analyzed (Participants) | 0

2. Primary Outcome: Number of Participants With Treatment Related Dose Delay or Treatment Discontinuation
Description: Adverse events will be recorded in relation to each cycle of treatment and graded according to CTCAE criteria. The toxicity co-primary outcome measure for the trial is defined as the occurrence of a treatment-related dose delay or treatment discontinuation due to toxicity
Time Frame: Through study completion, up to a maximum of 12 months. Serious AEs: Up to 90 days after last dose of study treatment, Other AEs: Up to 30 days after last dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Ramucirumab
Number analyzed (Participants) | 3
Participants | 3

ADVERSE EVENTS:
Time Frame: Up to a maximum of 12 months. Serious AEs: Up to 90 days after last dose of study treatment, Other AEs: Up to 30 days after last dose of study treatment
Arm/Group | Ramucirumab
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 3/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (N=3)
Neutropenic fever (Infections and infestations) | 1 (1)
pneumonia (Infections and infestations) | 2 (3)
bronchial occlusion (Respiratory, thoracic and mediastinal disorders) | 1 (2)
respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ramucirumab (N=3)
anemia (Blood and lymphatic system disorders) | 2 (10)
neutrophil count decreased (Blood and lymphatic system disorders) | 3 (4)
thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
leukocytosis (Blood and lymphatic system disorders) | 2 (2)
atrial fibrillation (Cardiac disorders) | 1 (1)
sinus tachycardia (Cardiac disorders) | 2 (3)
bradycardia (Cardiac disorders) | 1 (1)
dry eyes (Eye disorders) | 1 (1)
watery eyes (Eye disorders) | 1 (1)
eye redness (Eye disorders) | 1 (1)
abdominal pain (Gastrointestinal disorders) | 1 (2)
constipation (Gastrointestinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 1 (1)
clostridium difficile colitis (Infections and infestations) | 1 (1)
nausea and vomiting (Gastrointestinal disorders) | 1 (3)
fatigue (General disorders) | 3 (4)
hemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
pneumonia (Infections and infestations) | 1 (1)
shortness of breath (Respiratory, thoracic and mediastinal disorders) | 1 (2)
epistaxis (Blood and lymphatic system disorders) | 1 (2)
hyponatremia (Metabolism and nutrition disorders) | 1 (1)
hypocalcemia (Metabolism and nutrition disorders) | 1 (1)
hyperkalemia (Metabolism and nutrition disorders) | 1 (1)
anorexia (Metabolism and nutrition disorders) | 2 (4)
elevated creatinine (Renal and urinary disorders) | 1 (2)
acidosis (Metabolism and nutrition disorders) | 2 (2)
hematuria (Renal and urinary disorders) | 1 (1)
myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
hypotension (Cardiac disorders) | 2 (2)
hypertension (Cardiac disorders) | 1 (3)
mucositis (Gastrointestinal disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/08/NCT03904108/Prot_SAP_000.pdf